CLINICAL TRIAL: NCT05084599
Title: Effect of 90% Effective Dose of Metaraminol in Supine and Left Tilt Positions on Cesarean Section：A Non-inferiority Trial
Brief Title: Effect of 90% Effective Dose of Metaraminol in Supine and Left Tilt Positions on Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Head of Anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021PHB455-001
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Metaraminol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left-tilt group (Placebo Comparator): After spinal anesthesia, the patient was placed in a 15° left position until the fetus was delivered, and metaraminol was given at an initial rate of 2.00μg/kg/min throughout the process.
  Interventions: Drug: Metaraminol 2μg/kg/min
- supine group (Experimental): After spinal anesthesia, the patient was placed in a supine position until the fetus was delivered, and metaraminol was given at an initial rate of 2.7μg/kg/min throughout the process.
  Interventions: Drug: Metaraminol 2.7μg/kg/min

INTERVENTIONS:
Drug: Metaraminol 2.7μg/kg/min — After spinal anesthesia, the patient was placed in a supine position until the fetus was delivered, and metaraminol was given at an initial rate of 2.7μg/kg/min throughout the process.
  Arms: supine group
Drug: Metaraminol 2μg/kg/min — After spinal anesthesia, the patient was placed in left-tilt position until the fetus was delivered, and metaraminol was given at an initial rate of 2μg/kg/min throughout the process.
  Arms: left-tilt group

SUMMARY:
For hypotension after spinal anesthesia, metaraminol has different 90% effective doses in the supine position and the left-tilt position. We plan to conduct a non-inferiority trial to compare the effects of the two on the fetus and the mother.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy at term scheduled to be delivered via elective cesarean delivery;
2. height 150-180 cm;
3. American Society of Anesthesiologists (ASA) physical status II-III;
4. body mass index (BMI) <35 kg/m2.

Exclusion Criteria:

1. transverse presentation, fetal macrosomia;
2. uterine abnormalities (eg, large fibroids, bicornuate uterus);
3. polyhydramnios;
4. ruptured membranes, oligohydramnios;
5. intrauterine growth restriction;
6. gestational or nongestational hypertension, diabetes, or eclampsia;
7. hypertensive disorders or any condition associated with autonomic neuropathy (such as diabetes mellitus for >10 years) or renal failure;
8. contraindications for combined spinal-epidural anesthesia;
9. participants who declined to sign informed consent forms.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Umbilical artery blood pH | 30 seconds after delivery
  pH value of fetal umbilical artery blood

SECONDARY OUTCOMES:
hypotension | Intraoperative
  Number of Participants with systolic blood pressure reduction >20% baseline value or systolic blood pressure <90 mm Hg before delivery
bradycardia | Intraoperative
  Number of Participants with heart rate was ≤50 bpm before delivery Number of Participants with heart rate was ≤50 bpm before delivery Number of Participants with heart rate was ≤50 bpm before delivery
The incidence of nausea in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation.
Umbilical artery blood base excess | 30sec after delivery
  base excess of fetal umbilical artery blood
The incidence of vomiting in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yi, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes